CLINICAL TRIAL: NCT04283266
Title: Impact of a Synbiotic Containing Fructo-oligosaccharides and Bifidobacteria on Stool Frequency and Biological Markers in Middle-aged Adults: a Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Impact of a Synbiotic Containing Fructo-oligosaccharides and Bifidobacteria in Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vesale Pharmaceutica (Industry)
Collaborators: Université Catholique de Louvain (Other); University of Liege (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VesalePharma
Record Dates: First submitted 2019-11-12; First posted 2020-02-25 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Constipation
Keywords: probiotics; constipation; FOS
MeSH Terms: conditions — Constipation | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic group (Active Comparator): The synbiotic was composed of fructo-oligosaccharides (FOS): 4.95 g/ sachet and Bifidobacterium animalis lactis: 5 billion / sachet (n=13)
  Interventions: Dietary Supplement: Synbiotic
- Placebo group (Placebo Comparator): A placebo was composed of maltodextrin (60%) and sucrose (40%) : 5 g /sachet (n =14)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — Middle-aged subjects, who met ROME III criteria for constipation, received daily two sachets of synbiotic (Bifidobaterium animalis lactis Vesalius 002 and Fructo-Oligosaccharrides) for 5 days, then they received daily 1 sachet for the next 25 days
  Arms: Synbiotic group
Dietary Supplement: Placebo — Middle-aged subjects, who met ROME III criteria for constipation, received daily two sachets of placebo (maltodextrin and sucrose) for 5 days, then they received daily 1 sachet for the next 25 days
  Arms: Placebo group

SUMMARY:
The aim of the study is to evaluate the impact of a synbiotic containing fructo-oligosaccharides (FOS) and Bifidobacteria (VES002 LMG P-28149) on intestinal transit in middle-aged subjects characterized by a low number of defecations per week.

DETAILED DESCRIPTION:
Middle-aged subjects, who met ROME III criteria for constipation, received daily two sachets of either synbiotic or for 5 days, then they received daily 1 sachet for the next 25 days.

The primary endpoint of this trial is to evaluate the effect of supplementation in synbiotic containing fructo-oligosaccharides (FOS) and Bifidobacteria (VES002 LMG P-28149) on intestinal transit in middle-aged subjects characterized by a few bowel movements per week. The secondary endpoints are to evaluate both clinical criteria such as changes in stool appearance, quality of life and mood, relief and satisfaction of participants; and biological criteria such as changes in markers of gut function, low-grade chronic inflammation markers and gut microbiota composition. The safety of product use and compliance are also evaluated

Synbiotic group. The dietary supplement under study was composed of fructo-oligosaccharides - FOS: 4.95 gr / sachet and Bifidobacterium animalis lactis: VES002 (LMG P-28149): 5 billion / sachet. Sachets of powder were diluted in a in 200 ml of water at room temperature to be taken before breakfast. Doses were 2 sachets per day for the first 5 days and then 1 sachet per day for the next 25 days.

Placebo group. The placebo looked strictly identical to the synbiotic and contained only excipients (60% maltodextrin / 40% sucrose). Sachets of powder were diluted in a in 200 ml of water at room temperature to be taken before breakfast. Doses were 2 sachets per day for the first 5 days and then 1 sachet per day for the next 25 days.

ELIGIBILITY:
Inclusion Criteria:

* Free and informed consent
* Healthy male and female aged 50-70 years
* Patient with ≥1 and ≤3 bowel movements per week in the month before the selection visit and in the two weeks before the enrolment visit.
* At least one in four bowel movements had to involve hard faeces or separate lumps of faeces (Bristol scale class 1 in the three months before enrolment).

Exclusion Criteria:

* Subjects who, in the 30 days before the selection visit or at the time of the visit, had taken drugs, dietary supplements or any foodstuff enhanced in or containing substances, bacteria or yeasts that might have an effect on primary and secondary outcomes.
* Such products were also prohibited throughout the study.
* Subjects on a particular diet or who were under medical treatment that in the investigator's viewpoint might interfere with the evaluation of the study criteria
* Subjects who drink more than three glasses of wine a day or two 25 cl glasses of beer a day, or one glass of spirits per day.
* Subjects who drink more than five cups of coffee per day;
* Subjects with a body mass index (BMI) of more than 30,
* Subjects with type I or II diabetes,
* Subjects with constipation attributable to an organic or anatomical cause;
* Subjects with a history of chronic or inflammatory gastro-intestinal disease;
* Subjects with a history of digestive tract operation including bariatric surgery;

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-06-12 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
intestinal transit | daily evaluation (day-14 to day 30)
  stool frequency and consistency were investigated through daily self-assessment using the Bristol Stool Form Scale (BSFS). The BSFS classifies stools into 7 categories, including type 1, separate hard lumps, like nuts; type 2, sausage-shaped, but lumpy; type 3, like a sausage but with cracks on the surface; type 4, like a sausage or snake, smooth and soft; type 5, soft blobs with clear-cut edges; type 6, fluffy pieces with ragged edges, a mushy stool; type 7, watery, no solid pieces

SECONDARY OUTCOMES:
stool consistency | daily evaluation (day-14 to day 30)
  self-assessment using the Bristol Stool Form Scale
evaluation of quality of life | day 0 and day 30
  Mental and physical wellbeing were assessed before (d-14) and after intervention (d30) through the Short-Form 12-item (SF-12) questionnaire consisting of 12 questions relating to: physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations and general mental health (psychological distress and psychological well-being)
mood | daily evaluation (day-14 to day 30)
  Mood alterations was investigated through daily self-assessment using the Brief Mood Introspection Scale (BMIS), consisting of 16 mood adjectives (Lively, Drowsy, Happy, Grouchy, Sad, Peppy, Tired, Nervous, Caring, Calm, Content, Loving, Gloomy, fed up, Jittery, Active)47. Subjects were asked to circle the phrases describing their present mood (with XX = definitely do not feel; X = do not feel; V = slightly feel; VV = definitely feel on the diverse adjectives).
abdominal pain and intestinal discomfort | day -14 and day 30
  Evaluation based on VAS ( 0 - 100mm). 0 for no pain and 100 for unbearable pain
plasma inflammatory markers (pg/ml) | day 0 and day 30
  Plasma cytokines (interleukin (IL)-1alpha, IL-6, IL-8, IL-10, IL-17a, monocyte chemotactic protein-1 (MCP-1), interferon (IFN) gamma and tumor necrosis factor (TNF) alpha) measured by multiplex immunoassay (Millipore, Belgium) using Luminex® xMap® technology (Biorad, Nazareth, Belgium)
plasma gut peptides (pg/ml) | day 0 and day 30
  pancreatic polypeptide (PP), glucose-dependent insulinotropic peptide (GIP), leptin, ghrelin measured by multiplex immunoassay (Millipore, Belgium) using Luminex® xMap® technology (Biorad, Nazareth, Belgium)
microbiota composition | day 0 and day 30
  16S rDNA profiling, targeting V1-V3 hypervariable region and sequenced on Illumina MiSeq

IPD SHARING:
Plan to Share IPD: No